CLINICAL TRIAL: NCT06335940
Title: Admission for Respiratory Disease And VIdeo Regulation System
Acronym: ARAVIS-PED
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC23.0376
Record Dates: First submitted 2024-03-14; First posted 2024-03-28 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Pediatric Respiratory Diseases
Keywords: Videoregulation; Dispatch

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No videoregulation: An initial period of 40 days during which we leave the use of video-regulation to the discretion of the regulating physicians (emergency physicians or general practitioners) when they are faced with a call labelled by a medical regulation assistant (ARM) "Pediatric dyspnea in a child under 10 years of age" or when they themselves judge that the call falls into this category; as is the case in the current practice of the SAMU38.
- Videoregulation: A 40-day period during which we will encourage regulating physicians to use video-regulation for every call concerning "pediatric dyspnea in a child aged < 10 years".
  Interventions: Other: Videoregulation

INTERVENTIONS:
Other: Videoregulation — To encourage the use of video-regulation, several measures will be taken to reinforce its use as much as possible:
  * Posters visible to all in the dispatch room.
  * Regular mailings to all dispatching physicians.
  * On-site presence of interns and the study investigator to help doctors who are not used to video-regulation to get to grips with the computer tool.
  * Involvement of ARMs to remind doctors to use video-regulation.
  Groups: Videoregulation

SUMMARY:
Pediatric dyspnea is a major health problem, accounting for up to 27% of admissions to emergency departments in winter. It is estimated that a significant number (13%) of patients presenting to emergency departments are outpatients, at a time when emergency departments are having to cope with an ever-increasing flow of patients.

Proper referral of patients calling the SAMU Centre-15 takes on its full meaning in this context, but regulating paediatric calls is more difficult. Indeed, the regulating doctor is most often in contact with the parents, who describe what they see and pass on their concerns, and it is difficult to have direct contact with patients who are often very young. Obtaining objective criteria such as saturation and respiratory rate is also a real challenge.

To overcome the complexity of medical regulation, a number of tools and aids have been developed, including visio or video-regulation (regulation via the camera on the caller's smartphone).

This device has been evaluated in a number of situations, enabling it to take its place in the daily practice of many doctors, but there is very little data concerning pediatric visio-regulation, particularly with regard to dyspnea.

To the best of the investigator knowledge, there is no prospective study looking at the impact of Video-Regulation on the outcome of patients requiring the advice of SAMU Centre-15 for pediatric dyspnea.

ELIGIBILITY:
Inclusion Criteria:

* Age strictly less than 10 years
* Applicant calling the SAMU38 for a child with dyspnea announced or presumed by the interrogation.
* Patients for whom no opposition from parents has been obtained.
* Patients affiliated to social security

Exclusion Criteria:

* Call to organize a secondary intervention (or Inter-Hospital Transfer (TIH/TIIH)).
* Unsuccessful call (hung up when the dispatcher took the call, without the possibility of medical regulation).
* Refusal to take charge on arrival of rescue vector
* Call-back for a patient with an initial call to SAMU38 < 48h
* Means engaged by the CTA or an ARM even before medical regulation.

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients included in this study will be children strictly under 10 years of age whose parents have called the SAMU38 for respiratory difficulties.
  Therefore, patients who received ambulatory medical advice (with or without instructions to consult a general practitioner within a defined period of time), who were referred to the emergency service by their own means or who benefited from a first-aid vector (fire department or private ambulance) will be included.
Sampling Method: Non-Probability Sample
Enrollment: 588 (Estimated)
Dates: Start 2024-04-08 (Estimated); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-10-18 (Estimated)

PRIMARY OUTCOMES:
To determine in children under 10 years of age for whom a call to the SAMU38 for dyspnea is made, whether the use of Visio-Regulation reduces the percentage of emergency room admissions compared with standard telephone medical regulation. | 24 hours
  Percentage of participants with computerized admission to pediatric emergency departments

SECONDARY OUTCOMES:
Evaluate whether the use of video-regulation has an impact on the dispatcher's referral decision between ambulatory medicine and the emergency department. | through call completion, an average of 5 minutes
  Percentage of participants among all calls referred to outpatient and inpatient medicine
Determine whether the use of video-regulation leads to an increase in call time with the regulating doctor | through call completion, an average of 5 minutes
  Call time spent with the regulating physician
Evaluate parents' satisfaction with videoregulation compared with a standard call | 15 days
  Rating of appellants' satisfaction with the decision on a numerical scale from 1 to 5. 1 being the lowest level of satisfaction and 5 being the highest.
Evaluate the number of rescue vectors (fire brigade, private ambulance) triggered but whose decision will ultimately be to "leave on the spot" after the rescue worker's assessment. | through out-of-hospital care completion, an average of 1 hour
  Number of people left behind after a rescue vehicle has been deployed.
Evaluate whether the increased use of video-regulation is not associated with a higher rate of hospitalization in a conventional ward or intensive care unit | 24 hours
  Number of patients admitted to hospital or intensive care/resuscitation after emergency admission within 24 hours of the call